CLINICAL TRIAL: NCT05470842
Title: How Common is Hypoglycaemia in Older People With Diabetes Who Have Falls, Dizziness or Other Symptoms Suggestive of Hypoglycaemia? A Continuous Glucose Monitoring Study
Brief Title: How Common is Hypoglycaemia in Older People With Diabetes Who Fall?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: v2
Record Dates: First submitted 2022-07-19; First posted 2022-07-22 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2023-11

CONDITIONS: Diabetes; Hypoglycaemia
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: Single-centre, single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Continuous glucose monitoring (Experimental): Continuous Glucose Monitoring Device for up to 10 days
  Interventions: Device: Continuous glucose monitoring (Dexcom G6)

INTERVENTIONS:
Device: Continuous glucose monitoring (Dexcom G6) — All participants will be issued with the Dexcom G6 device. The trial team will buy the readers or smartphones and sensors and provide the participants with all the necessary equipment. Participants will be shown how to wear the Dexcom G6 device, which they will be asked to wear for up to 10 days (=the lifespan of one sensor).
  There will be no change in the standard care of the participants' diabetes management, during the study period.
  Other Names: Dexcom G6

SUMMARY:
The purpose of this study is to use 24 hour continuous glucose monitoring in older patients with diabetes who present with symptoms of falls, or dizziness, or confusion, that may indicate hypoglycaemia.

DETAILED DESCRIPTION:
Background and study aims Patients with diabetes can be treated with medications (such as insulin or sulfonylureas) that can lower the sugar levels too much (hypos). A hypo means that the brain does not get enough energy. A person can become confused, dizzy, pass out, and/or have a fall.

Older people with diabetes often seek treatment in hospital for symptoms such as falls, dizziness or feeling muddled. Health care professionals will order tests to investigate the possible causes for the fall, being muddled or dizzy, which can include a review of medications, checking blood pressures and the heart.

However, it has previously been difficult to obtain 24-hour blood sugar monitoring in older people with diabetes to check if hypos could be an important contributing factor to their falls and dizzy spells.

Continuous Glucose Monitoring (CGM) allows non-stop monitoring with a sensor that sits just under the skin. This sends sugar readings to a smartphone every few minutes (via Bluetooth) for 10 days. This enables full evaluation of the amount of time a person's sugar is in the target range, and the time in the low/high ranges. Medical research with CGM has revealed that some older people are suffering from substantial periods of hypos that they are not aware of.

During this study, older people with diabetes will be asked to wear a CGM device for 10 days to investigate possibility of hypos.

ELIGIBILITY:
Inclusion Criteria:

* 75 years and older with diabetes
* Treated with glucose-medications which carry a high risk of hypoglycaemia (sulfonylureas and/or insulin)
* Presenting to hospital with a fall and/or symptoms suggestive of unrecognised hypoglycaemia (such as dizziness, feeling muddled).

Exclusion Criteria:

* Treatment with metformin alone
* Lack of capacity,
* Not willing to participate,
* Terminal illness (less than one-year life expectancy).
* Evidence of bruising, bleeding, cellulitis and/or skin tears on the upper arms or abdomen.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Mattishent, PhD, Principal Investigator — University of East Anglia
Locations (1):
- University of East Anglia, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Glucose Monitoring: Continuous Glucose Monitoring Device for up to 10 days
  Continuous glucose monitoring (Dexcom G6): All participants will be issued with the Dexcom G6 device. The trial team will buy the readers or smartphones and sensors and provide the participants with all the necessary equipment. Participants will be shown how to wear the Dexcom G6 device, which they will be asked to wear for up to 10 days (=the lifespan of one sensor).
  There will be no change in the standard care of the participants' diabetes management, during the study period.
Period: Overall Study
Arm/Group | Continuous Glucose Monitoring
Started | 12
Completed | 11
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Continuous Glucose Monitoring
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Captured Hypoglycaemia
Description: Number of patients who experienced more than 15 minutes of hypoglycaemia within the 10-day sensor lifespan and data capture period.
Time Frame: 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitoring
Number analyzed (Participants) | 11
Participants | 3

2. Secondary Outcome: Overall Time in Range (Average)
Description: The percentage of time glucose concentrations in the 10-day monitoring period that were within the defined target range (3.9 - 10.0 mmol) as specified by international consensus.
Time Frame: 10 days
Population: Completers of the monitoring period
Measure: Mean (Standard Deviation); unit: percentage of Time in Range
Arm/Group | Continuous Glucose Monitoring
Number analyzed (Participants) | 11
percentage of Time in Range | 52 (23)

3. Secondary Outcome: Emergency Department Re-attendances and/or Hospital Re-admissions for Falls, Fractures, Heart Attacks, Ischaemic Strokes and Death Within 30 Days
Description: Number of participants with hospital admissions and emergency department attendances within 30 days of sensor monitoring. Review of hospital records to ascertain date of admission and clinical presentation.
Time Frame: 30 days
Population: Completers analysed
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitoring
Number analyzed (Participants) | 11
Participants | 1

4. Other Pre Specified Outcome: For Participants Who Experienced Hypoglycaemic Events, the Amount of Time (Minutes) They Were in the Hypoglycaemic Range
Description: Number of minutes the blood glucose was within the hypoglycaemic range in the participants who experienced hypoglycaemic events.
Time Frame: 10 days
Population: Subgroup of participants who were found to have hypoglycaemic events
Measure: Median (Full Range); unit: minutes
Arm/Group | Continuous Glucose Monitoring
Number analyzed (Participants) | 3
minutes | 40 [30 to 330]

ADVERSE EVENTS:
Time Frame: 30 days from completion of collection of continuous glucose monitoring data
Arm/Group | Continuous Glucose Monitoring
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Continuous Glucose Monitoring (N=11)
Congestive cardiac failure (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT05470842/Prot_SAP_000.pdf